CLINICAL TRIAL: NCT07024030
Title: A Clinical Phase I/II Study Evaluating the Safety, Tolerability and Pharmacokinetics of the PSMA-targeted Fluorescent Contrast Agent DGPR1008 for Intraoperative Imaging in Prostate Cancer
Brief Title: Safety and Efficacy Trial of a Targeted PSMA Fluorescent Contrast Agent (DGPR1008) for Intraoperative Imaging of Prostate Cancer
Acronym: DGPR1008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haitao Niu, MD (Other)
Responsible Party: Sponsor-Investigator, Haitao Niu, MD, Member of the Standing Committee of the Party Committee, Vice President of Qingdao University,, The Affiliated Hospital of Qingdao University
Organization: The Affiliated Hospital of Qingdao University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2024-047-04; CXHL2400243 (Other: NMPA)
Record Dates: First submitted 2025-05-18; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy
Keywords: DGPR1008
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The first dose group (Experimental): Slowly infuse intravenously 24 hours before the scheduled surgery. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Interventions: Drug: 0.02mg/kg
- The second dose group (Experimental): Slowly infuse intravenously 24 hours before the scheduled surgery. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Interventions: Drug: 0.04mg/kg

INTERVENTIONS:
Drug: 0.02mg/kg — Slowly infuse intravenously 24 hours before the scheduled surgery. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Other Names: intravenous drip
  Arms: The first dose group
Drug: 0.04mg/kg — Slowly infuse intravenously 24 hours before the scheduled surgery. The investigator shall conduct near-infrared fluorescence imaging during the operation to assist with the surgery. Tissues detected with fluorescence need to be marked, and resection shall be guided by fluorescence until there is no fluorescent tissue within the surgical field.
  Other Names: intravenous drip
  Arms: The second dose group

SUMMARY:
a single-arm, open-label, multi-center study to evaluate safety, tolerability, pharmacokinetics, and the effectiveness of near-infrared fluorescence imaging during surgery.

DETAILED DESCRIPTION:
We plan to enroll 24 prostate cancer patients and divide them into 2 dosage groups. Intravenous administration will be conducted 24 hours before surgery. Blood samples will be collected for relevant tests, and fluorescence imaging will be performed during the operation. After surgery, the intraoperative imaging results will be compared with pathological findings to draw relevant conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide informed consent prior to enrollment, fully understand the trial details, adverse events, and communicate effectively with investigators. Written informed consent must be voluntarily signed.

Adult male subjects aged ≥18 years. Subjects with pathologically confirmed prostate cancer (Gleason score ≥7) via pre - operative prostate biopsy, scheduled for radical prostatectomy.

No significant liver or kidney impairment: liver - total bilirubin ≤2×ULN (except Gilbert syndrome), ALT/AST ≤3×ULN; kidney - creatinine clearance rate ≥50 mL/min/1.73m² (simplified MDRD).

No surgical contraindications; suitable for laparoscopic radical prostatectomy as determined by the investigator.

Subject and partner/spouse agree to avoid conception and sperm donation from screening until 3 months post - trial, and use effective contraception.

Exclusion Criteria:

* Subjects will be excluded if any of the following apply:

Allergic constitution (history of allergy to ≥2 drugs), prone to allergic reactions, or allergic to the investigational drug (including components).

Clinically significant abnormal screening results affecting the study, or serious concomitant diseases (except stable cases approved by the investigator).

Participation in other clinical trials and received investigational products within 1 month before study drug administration.

Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of single-dose administration of DGPR1008 in patients | From the screening period to the day before withdrawal on Day 3 of the trial
  Adverse event collection, including (such as the location, nature, and frequency of pain), physical signs (such as the scope of rash, blood pressure values), laboratory abnormal values and units (such as ALT 200 U/L), etc.
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the area under the plasma concentration-time curve from time 0 to infinity (AUC₀-∞) in the blood of 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the maximum plasma concentration (Cmax) in the blood of 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the area under the plasma concentration-time curve from time 0 to time t (AUC₀-t) in the blood of 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the percentage of extrapolated area under the plasma concentration-time curve (AUC%Extrap) in the blood of 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the plasma elimination half-life (t₁/₂) in 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the blood clearance (CL) in 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the renal clearance (CL renal) in 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the terminal elimination rate constant (λz) in 24 subjects
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the apparent volume of distribution during terminal phase (Vz) in 24 subjects
To evaluate the safety of single-dose administration of DGPR1008 in patients | From the screening period to the day before withdrawal on Day 3 of the trial
  Vital signs examination, such as blood pressure, oxygen saturation, pulse and other data.
To evaluate the pharmacokinetic characteristics of single-dose administration of DGPR1008 in patients | PK blood samples will be collected 60 minutes before drug administration, and immediately, 30 minutes (±5 minutes), 1 hour (±10 minutes), 2 hours (±10 minutes), 4 hours (±20 minutes), 6 hours (±30 minutes), and 8 hours (±30 minutes) after administration.
  To measure the mean residence time (MRT₀-t, MRT₀-∞) of the drug in the blood of 24 subjects
To evaluate the safety of single-dose administration of DGPR1008 in patients | From the screening period to the day before withdrawal on Day 3 of the trial
  Physical examination, with body mass index (BMI) reported as weight (kg)/height (m²), electrocardiogram (ECG) examination, and laboratory tests (blood routine, blood biochemistry, urinalysis, coagulation function).

SECONDARY OUTCOMES:
Evaluate the effectiveness of the detection by DGPR1008 in conjunction with the near-infrared fluorescence imaging device for intraoperative imaging in patients. | 24 hours before the surgery
  Evaluate the sensitivity, specificity, false positive rate, false negative rate of DGPR1008 in detecting prostate cancer cells or tissues in near-infrared imaging, and assess the tumor-to-background ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided